CLINICAL TRIAL: NCT06592352
Title: MODAFIMS: An Open-label, Single-center Clinical Trial to Evaluate Predictors of Response to MODAFinil in the Treatment of Cognitive Deficits in Patients With Multiple Sclerosis
Brief Title: MODAFIMS: A Trial to Evaluate Predictors of Response to MODAFinil in Patients With Multiple Sclerosis
Acronym: MODAFIMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MODAFIMS; 2022-501414-53-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-03; First posted 2024-09-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: multiple sclerosis; cognitive impairment; functional MRI
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: single-center, open-label design to evaluate the effect of modafinil on cognitive deficits in adult patients with multiple sclerosis and identify predictors of response using functional Magnetic Resonance Imaging (fMRI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modafinil Generis 100 mg (Experimental): Modafinil Generis 100 mg, in a dose of 200mg, once a day, orally.
  Interventions: Drug: Modafinil Generis 100 mg

INTERVENTIONS:
Drug: Modafinil Generis 100 mg — All participants enrolled in the study will receive the study intervention drug (Modafinil Generis 100 mg). Dose 200 mg once per day (2 tablets of 100 mg) in the morning for 3 months (84 days), Oral administration
  Other Names: Modafinil Generis

SUMMARY:
This is a phase II/exploratory clinical trial with a single-center, open-label design to evaluate the effect of modafinil on cognitive deficits in adult patients with multiple sclerosis and identify predictors of response using functional Magnetic Resonance Imaging (fMRI).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a neurodegenerative disease that affects the central nervous system. There are no commercially authorized therapeutic options available for the treatment of cognitive impairment in patients with multiple sclerosis. It is then necessary to conduct robust clinical trials to select better therapies.

Modafinil is a drug approved by INFARMED and European Medicines Agency (EMA) for the treatment of excessive sleepiness associated with narcolepsy. Modafinil has been tested in 5 clinical trials in patients with multiple sclerosis and the results indicated a potential improvement in cognitive deficits in tasks that measure executive function, verbal memory, and/or working memory performance.

Despite encouraging results, there is a huge variation in its effect in individual patients and a significant proportion of sub-optimal/non-responders. Therefore, it is important to identify personalized predictors of response to best tailor the treatment to each patient.

This is a phase II/exploratory clinical trial with a single-center, open-label design to evaluate the effect of modafinil on cognitive deficits in adult patients with multiple sclerosis and identify predictors of response using functional Magnetic Resonance Imaging (fMRI).

The primary objective of the clinical trial is to identify fMRI markers of response to modafinil. In other words, our aim is to analyse brain activity (using fMRI) before and after modafinil intake and select the features that can better differentiate between responders and non-responders. These patient groups will be determined according to the improvement rate in the Symbol digit modalities test (SDMT) - which will be evaluated at screening, baseline and at the end of treatment.

The clinical trial will be conducted at Centro Clínico Académico - Braga, Associação (2CA-Braga), Unidade Local de Saúde de Braga (ULS Braga), E.P.E.. Participants will be recruited at the outpatient unit of the Neurology department of ULS de Braga.

A total of 64 eligible patients will be enrolled to receive modafinil at a dose 200 mg (2 tablets of 100 mg) once per day in the morning for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for the participation in the trial.
* Patients that are able to read and write.
* Male or female, aged between 18 and 64 years old at the time of signing the ICF.
* Diagnosed with Relapsing-Remitting MS or Clinically Isolated Syndrome, according to McDonald 2017 diagnostic criteria (Thompson et al., 2018).
* Expanded disability status score (EDSS) less than 6.5.
* Presence of subjective cognitive complaints.
* SDMT score (number of correct responses within 90 seconds) at Screening ≤ 55 (Benedict et al., 2016; Parmenter et al., 2007).
* Female participants of childbearing potential and male participants whose partner is of childbearing potential must be willing to ensure that they or their partner use protocol's recommended effective contraception methods, which is not based only on hormonal methods, during all the 6 months of the trial (3 months of treatment plus 3 months of safety follow-up).
* Male participants must agree to refrain from donation of semen from first study treatment administration up to at least 90 days after last administration.
* Participants, that in the medical investigator's opinion, are able and willing to comply with all trial requirements.

Exclusion Criteria:

* Female participant who is pregnant, breastfeeding or planning pregnancy during the trial.
* Participants who have participated in another research trial involving an investigational product within the past 5 half-lives of the other investigational product.
* Participants who have any disability that, in the opinion of the investigator, significantly interferes with the neuropsychological testing and/or the tasks in the functional MRI.
* Participants not able to undergo MRI scanning.
* Participants who have any contra-indication for taking modafinil, according to the prescribing information and SmPC, such as hypersensitivity to the active substance and any excipient present in the modafinil or any documented adverse reaction after modafinil intake.
* Participants with known hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Participants with a history of left ventricular hypertrophy or cor pulmonale and patients with mitral valve prolapse who developed mitral valve prolapse syndrome when previously treated with central nervous system stimulants.
* Current use of modafinil, armodafinil.
* Current use of other psychostimulants, including amphetamines, cocaine, bupropion, gingko biloba, among others, and beverages or food containing methylxanthines (e.g., coffee, tea, cola, caffeine, chocolate, sodas) exceeding 500 mg methylxanthines per day (for example, consumption of more than 5 espresso coffees or 100 mg of dark chocolate per day; Sanchez, 2017).
* Significant neurological history aside from MS (e.g., Epilepsy).
* Significant psychiatric history (e.g., Schizophrenia, Bipolar Disorder, Major Depression, severe anxiety disorder, aggressive or hostile behaviour).
* A documented history of attempted suicide in the last 2 years OR suicidal ideation with intent, with or without a plan or method (e.g., positive response to items 4 or 5 in the assessment of suicidal ideation on the C-SSRS) over the 6 months prior to the Screening Visit.
* Significant insomnia (grade > 1 according to Common Terminology Criteria for Adverse Events, CTCAE v5)
* History of severe hypersensitivity reactions to any medicine.
* Presence of any clinically significant abnormality in ECG morphology or ECG parameters.
* Known immunodeficiency syndrome.
* Have serum alanine aminotransferase (ALT) values greater than 3 times the upper limit of normal at screening.
* Positive test for anti-Human Immunodeficiency virus 1 or 2 antibodies, Hepatitis B surface antigen (HBsAg) or anti Hepatitis C virus antibodies.
* Creatinine clearance < 20 ml/min determined by Cockcroft-Gault equation.
* History of alcoholism or drug abuse.
* Average daily consumption of more than 20 cigarettes.
* Participants with disability that interferes with the performance of the CT procedures (for example, motor deficit in upper limb, decreased visual acuity even with correction).
* Participants with increased risk of epileptic seizures, history of cardiac arrhythmias, or uncontrolled moderate to severe hypertension.
* Participants taking warfarin or any other prohibited medication.
* Sleep complaints confirmed by Epworth Sleepiness Scale (ESS) scale score >10 at screening visit OR known sleep disorder.
* Any other condition that, in the opinion of the investigator, contra-indicates the participation of the patient.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Acute changes in brain fuction and connectivity measured using resting state fMRI. | Day 1 (baseline): before and 3 hours (± 30 minutes) after modafinil administration.
  Acute changes in brain functional connectivity at rest will be measured using resting-state fMRI through Echo-planar imaging (EPI) sequences.
Long-term changes in brain function and connectivity measured using resting state fMRI. | Day 1 (baseline), 3 hours (± 30 minutes) after medication; and Day 84 (3 months after treatment with modafinil), 3 hours (±30 minutes) after medication.
  Long-term changes inbrain functional connectivity at rest will be measured using resting-state fMRI through Echo-planar imaging (EPI) sequences.

SECONDARY OUTCOMES:
Acute changes in brain function and connectivity measured using a Go/no-Go task fMRI. | Baseline (day 1): before and 3 hours (± 30 minutes) after modafinil administration.
  Acute changes in brain activity during a Go/No-Go task, measured using task-based fMRI through Echo-planar imaging (EPI) sequences.
Long-term changes in brain function and connectivity measured using a Go/no-Go task fMRI. | Day 1 (baseline), 3 hours (± 30 minutes) after medication; and Day 84 (3 months after treatment with modafinil), 3 hours (±30 minutes) after medication.
  Long-term changes in brain activity during a Go/No-Go task, measured using task-based fMRI through Echo-planar imaging (EPI) sequences.
SDMT score | Day 1 (baseline) and Day 84 (3 months after treatment)
  Symbol Digit Modalities Test (SDMT) is a cognitive function test to assess visual attention and information processing speed, which involves a simple substitution task. The SDMT includes a reference key of 9 symbols, each paired with a single digit. Below the reference key are rows of symbols arranged randomly. The participant will have 90 seconds to say out loud the number that corresponds to each symbol. Answers are registered by the rater in the SDMT form and the score corresponds to the number of correct answers given within the 90-seconds interval. A decrease of 4 points from baseline on the SDMT is considered a meaningful worsening.
Stroop test | Screening and Day 84 (3 months after treatment)
  The Stroop test is a measure of executive function, including selective attention capacity, processing speed, behaviour inhibition and interference resistance. The performance in this test is measured by the interference index.
MS-QoL-54 total score | Screening and Day 84 (3 months after treatment).
  Multiple Sclerosis Quality of Life-54 (MS-QoL-54) is a multidimensional health-related quality of life (QoL) measure combining generic and MS-specific items into a single tool. MS-QoL-54 has a total of 54-items generating 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall QoL, and sexual function.
  The single item measures are satisfaction with sexual function and change in health. The summary scores are the physical health composite summary and the mental health composite summary. Scores range from 0 to 100, with higher values representing a better QoL.
WPAI:MS total score | Screening and Day 84 (3 months after treatment).
  The Work Productivity and Activity Impairment Questionnaire for MS is a 6-item questionnaire which measures the impact of MS on the patients' work productivity (including the duration of work time missed due to the disease and decrease in productivity when working while experiencing symptoms) and non-working activities (for example, childcare) during the past seven days.
MFIS total score | Screening and Day 84 (3 months after treatment).
  The Modified Fatigue Impact Scale (MFIS) is a 21-item tool used to rate the impact of fatigue during the last 4 weeks on a 5-point Likert scale, from "Never" (0) to "Almost always" (4). The total score is the sum of all items from 0 to 84, with higher scores indicating greater impact of fatigue.
PDQ total score | Screening and Day 84 (3 months after treatment with modafinil)
  Perceived Deficits Questionnaire (PDQ) is a 20-items self-report measure to assess perceived cognitive impairment during the past 4 weeks. The total score ranges from 0 to 80, and higher scores reflect greater perceived cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: João Cerqueira, MD, PhD, Principal Investigator — 2CA-Braga
Locations (1):
- Clinical Academic Center - Braga (2CA-Braga), Braga, Portugal

IPD SHARING:
Plan to Share IPD: No